CLINICAL TRIAL: NCT05522296
Title: Break-through Infection Following Mpox vaccinatIon: Target Trial Emulation
Brief Title: Break-through Infection Following Mpox vaccinatIon
Acronym: REMAIN
Status: Completed | Type: Observational
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: Department of Health, Generalitat de Catalunya (Other Government); Hospital Vall d'Hebron (Other); Hospital Clinic of Barcelona (Other); Hospital Universitario 12 de Octubre (Other); Public Health Service of Madrid (Other); Madrid Salud (Other); Harvard School of Public Health (HSPH) (Other); London School of Hygiene and Tropical Medicine (Other); Germans Trias i Pujol Hospital (Other); BCN Checkpoint (Industry); Centro de Saluld Sandoval (Unknown); Centro de Salud Montesa (Unknown); Hospital Nacional Arzobispo Loayza (Other); Hospital Regional III Honorio Delgado (Unknown); Hospital Regional Docente de Trujillo (Unknown); Instituto Conmemorativo Gorgas de Estudios de la Salud (Unknown); Ministerio de Salud de Panamá (Unknown); Fundación Arriaran (Unknown)
Responsible Party: Principal Investigator, Oriol Mitja, Associate Professor, Infectious Diseases and Global Health, Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia
Other Study IDs: REMAIN
Record Dates: First submitted 2022-08-27; First posted 2022-08-31 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Mpox
Keywords: Monkeypox; Mpox Vaccine; Intradermal Mpox vaccine; Mpox
MeSH Terms: conditions — Mpox, Monkeypox | interventions — Smallpox Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unvaccinated: Unvaccinated individuals who have risk factors for mpox infection and do not have a past history of mpox infection
- Vaccinated: Vaccinated individuals with smallpox and mpox vaccine (Live Modified Vaccinia Virus Ankara) who have risk factors for monkeypox infection and do not have a past history of mpox infection.
  Interventions: Drug: Mpox Vaccine

INTERVENTIONS:
Drug: Mpox Vaccine — Vaccination with smallpox and mpox vaccine (Live Modified Vaccinia Virus Ankara)
  Groups: Vaccinated

SUMMARY:
The purpose of this study is to assess the protection of smallpox preexposure vaccination against infection with mpox in real-world individuals with risk factors for mpox.

DETAILED DESCRIPTION:
A Target Trial Emulation study that tries to emulate the sequential specification of a target trial will be conducted measuring and controlling confounders when there is a common cause of vaccination and outcome event.

Participants will be provided with a Quick response (QR) code to access the RedCap study platform, which will guide them to the enrolment process. If the participant accepts and meets all the inclusion and none of the exclusion criteria, they will be directed to a baseline survey to self-collect sociodemographic data and information regarding risk factors, sexual behaviour, vaccination, and exposure to mpox.

Newly vaccinated participants will be matched 1:1 to unvaccinated controls. The matching will be performed based on the site of recruitment, and self-reported baseline sexual health and practices. Vaccinated and unvaccinated participants will be matched on variables associated with the probability of infection.

Follow-up will include regular surveys every month from the index date (i.e., enrolment date in the unvaccinated group, or vaccination date for the vaccinated group), to collect data on change on risk factors, sexual behaviour in the past month, vaccination status, and exposure to mpox. The participant will be asked to self-report if they develop symptoms suggestive of mpox, and the study platform will direct them to a specific mpox infection survey.

For each participant, follow-up will end at the earliest of the following events: mpox infection, voluntary withdraw, or the end of the study period. A health record review will be conducted to corroborate the diagnosis of new cases and to provide validity to the self-report.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 years or older.
2. Individuals with general risk factors for mpox infection, as currently defined by the local guidelines for vaccination. These risk factors include at least one of the following items:

   * Individual-reported use of HIV pre-exposure prophylaxis (PrEP).
   * Individual-reported chemsex practices
   * Individual-reported multiple sexual partners.
   * Individuals with a history of a sexually transmitted infection (STI) in the past year.
   * Individuals living with HIV infection.
3. Signature of informed consent.

Exclusion Criteria:

1. Unable to provide signature of informed consent.
2. Past infection with monkeypox.
3. Past smallpox vaccination.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male cis and Female trans
Study Population: Vaccinated and unvaccinated individuals who have risk factors for mpox infection and do not have a past history of mpox infection.
Sampling Method: Non-Probability Sample
Enrollment: 3125 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Polymerase chain reaction (PCR)-confirmed mpox infection | From 14 days after the index date to twelve months after the index date
  Mpox PCR positivity in participants with mpox infection symptoms

SECONDARY OUTCOMES:
Polymerase chain reaction (PCR)-confirmed mpox infection | From immediately after the index date to twelve months after the index date
  Mpox PCR positivity in participants with mpox infection symptoms
Duration of general symptoms | From 14 days after the index date to twelve months after the index date
  Time from onset to resolution of general symptoms in participants with PCR-confirmed mpox infection (in days).
Severity of rash | From 14 days after the index date to twelve months after the index date
  Number of mpox lesions (lesions count)
Duration of skin rash | From 14 days after the index date to twelve months after the index date
  Time from onset to resolution of skin rash in participants with PCR-confirmed
Medical treatment | From 14 days after the index date to twelve months after the index date
  Requirement of medical treatment (yes/no)
Hospitalization | From 14 days after the index date to twelve months after the index date
  Requirement of hospital admission (yes/no)
Scarring | From 14 days after the index date to twelve months after the index date
  Residual scarring after mpox (yes/no)
Safety and tolerability | One month after vaccination
  Description of systemic and skin reactions

CONTACTS AND LOCATIONS:
Locations (6):
- Hospital Clínico San Borja Arriarán, Santiago, Santiago Metropolitan, Chile
- Instituto Conmemorativo Gorgas de Estudios de la Salud (ICGES), Panama City, Panama
- Peru (3):
  - Hospital Regional III Honorio Delgado, Arequipa
  - Hospital Nacional Arzobispo Loayza, Lima
  - Hospital Regional Docente de Trujillo, Trujillo
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Upon request after publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After Publication

REFERENCES:
- [Background] Barda N, Dagan N, Ben-Shlomo Y, Kepten E, Waxman J, Ohana R, Hernan MA, Lipsitch M, Kohane I, Netzer D, Reis BY, Balicer RD. Safety of the BNT162b2 mRNA Covid-19 Vaccine in a Nationwide Setting. N Engl J Med. 2021 Sep 16;385(12):1078-1090. doi: 10.1056/NEJMoa2110475. Epub 2021 Aug 25. PMID 34432976
- See also: Recommendations of experts in trial design to World Health Organization — https://www.who.int/news-room/events/detail/2022/08/02/default-calendar/who-monkeypox-research---what-study-designs-can-be-used-to-address-the-remaining-knowledge-gaps-for-monkeypox-vaccines
- See also: Spanish incidence estimation document for the calculation of the number of participants — https://www.ema.europa.eu/en/news/emas-emergency-task-force-advises-intradermal-use-imvanex-jynneos-against-monkeypox